CLINICAL TRIAL: NCT02809742
Title: Intermittent Bolus Administration of Ropivacaine for Epidural Labor Analgesia : an Observational Study
Brief Title: Intermittent Ropivacaine Bolus for Epidural Labor Analgesia
Acronym: OptimEpi
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Philippe Cuvillon, MD, PhD, Centre Hospitalier Universitaire de Nīmes
Other Study IDs: PMCurrieU2
Record Dates: First submitted 2016-05-31; First posted 2016-06-22 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Labor Pain
Keywords: Pregnant; Labor; Epidural; Analgesia; Intermittent
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Epidural group: Epidural : automatic intermittent boluses ( 8-12 mL per hour) + patient controlled bolus (4 mL evrey 20 min) using ropivacaine
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Epidural : automatic intermittent boluses associated with patient controlled bolus using ropivacaine
  Other Names: ropivacaine 2 mg/ml

SUMMARY:
Enhanced patient safety and satisfaction have contributed to growing use of epidural labor analgesia. Epidural analgesia appears to be currently the most effective technique in reducing pain during labor. However, reduction in total dose of local anesthetic and thus motor blockade is crucial to improve the obstetric outcome. This technique has evolved from intermittent boluses by anesthesiologists to the current standard labor epidural analgesic regimens in many institutions in North America and Europe that consist of a local anesthetic in combination with an opioid delivered via continuous epidural infusion (CEI) with or without patient-controlled epidural analgesia (PCEA) boluses. Recently,a new mode of administration has been used: regular bolus of low concentration local anesthetic + intermittent bolus (PIEB). This technique would offer safe and superior quality labor analgesia and greater maternal satisfaction by reducing total amount of the drug combination.

The primary outcome was to evaluate the analgesic efficacy of PIEB epidural drug delivery in terms of visual analogue scale satisfaction (VAS) score in a large cohort of patients. The secondary outcomes were to measure the degree of motor blockade, neonatal and obstetric outcomes, total drug dose and incidence of pain that required top-up administration (breakthrough pain)

DETAILED DESCRIPTION:
Patients were explained about the procedure and written informed consent was obtained. Healthy term primi or second gravid parturients (aged >18 years) with a singleton, live fetus in vertex presentation when in active stage of labor with cervical dilation of 3-5 cm were recruited in the study after they requested epidural for pain relief. PIEB epidural analgesia was used.

Primary outcome was maternal satisfaction during labor and delivery. Our hypothesis was that patients would have a greater level of satisfaction when using PIEB technique. The secondary outcomes were to measure the degree of motor blockade, neonatal and obstetric outcomes.

ELIGIBILITY:
Inclusion Criteria:

* healthy term primi or second gravid parturients
* aged 18-30 years
* singleton, live fetus
* vertex presentation
* active stage of labor with cervical dilation of 3-5 cm parturients

Exclusion Criteria:

* Hypertension
* no vertex presentation
* contraindications to neuraxial blockade

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: healthy term primi or second gravid parturients aged 18-30 years with a singleton, live fetus in vertex presentation when in active stage of labor with cervical dilation of 3-5 cm
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Verbal Analogue Satisfaction Score | 1 day
  VASS: 0-10: 0 = no satisfaction to 10 (total satisfaction)

SECONDARY OUTCOMES:
maternal hypotension | 1 day
  Evaluation of adverse events over epidural infusion (mean arterial pressure< 65 mmHg)
Apgar score | 1 day
  The Apgar test is done by a doctor, midwife, or nurse. The health care provider examines the baby's:
  * Breathing effort
  * Heart rate
  * Muscle tone
  * Reflexes
  * Skin color
  Each category is scored with 0, 1, or 2, depending on the observed condition.
Anesthetic rescue | 1 day
  Evaluation of the rescue performed by anesthesist over infusion
nausea | 1 day
  Number of maternal nausea event
fetal heart rate | 1 day
  Fetal heart sounds were monitored with a continuous Doppler machine
Motor blockade | 1 day
  Bromage score for maternal motor block

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nimes, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No